CLINICAL TRIAL: NCT04207593
Title: Prospective, Randomized, Controlled Trial of the Effect of Long-term Oxygen Therapy on 6-minute Walking Distance, Clinical Parameters and Hemodynamics in Patients With PAH and CTEPH
Brief Title: The Effect of Oxygen Therapy on 6MWD in PAH and CTEPH Patients With Hypoxemia
Acronym: SOPHA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ekkehard Gruenig, Prof. Dr. med. Ekkehard Grünig; Head of centre for pulmonary hypertension, Thoraxklinik-Heidelberg gGmbH
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-11SO*
Record Dates: First submitted 2019-12-17; First posted 2019-12-23 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Oxygen Deficiency; Pulmonary Arterial Hypertension; CTEPH
Keywords: Oxygen; Pulmonary Arterial Hypertension; CTEPH; 6MWD
MeSH Terms: conditions — Hypoxia; Pulmonary Arterial Hypertension | interventions — Oxygen

STUDY DESIGN:
Masking Description: PAH patients experiencing oxygen desaturations at rest and during physical activity, when O2 partial pressure is repeatedly <8 kPa (<60 mmHg; alternatively, 90% of O2 saturation). Patients will be divided in a supplemental-oxygen group (primary intervention group) and no-supplemental-oxygen group (control group). Patients of the control group will be offered to participate in the interventional treatment arm after they have terminated the control period (partial cross-over; secondary intervention group). Randomization will be performed in a 1:1 ratio. Randomization to one of the groups will be performed by block randomization. Randomization lists will be created by the data management using a computer to generate random numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxygen Therapy provided (Active Comparator): Patients will be divided in a supplemental-oxygen group (primary intervention group) throughout the study
  Interventions: Drug: Oxygen
- no-supplemental-oxygen group (control group) (Sham Comparator): Patients of the control group will beginn the study without Oxygen Therapie and will be offered to participate in the interventional treatment arm after they have terminated the control period (partial cross-over; secondary intervention group).
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Study medication will be oxygen (O2) in diverse concentrations, titrated until a SaO2>90% or pO2 >60 mmHg is achieved, for 20 patients vs. no supplemental O2 for 20 patients over 90 ± 7 days. Patients of the control group will be offered to participate in the interventional treatment arm after they have terminated the control period (partial cross-over; secondary intervention group). After the end of the study it is up to the judgment of the investigator to prescribe oxygen to all patients who might benefit from the treatment.
  Other Names: Liquid oxygen

SUMMARY:
Treatment of O2 naïve patients with PAH will be included in this investigator-initiated trial (IIT) to assess efficacy and safety of oxygen substitution. Nocturnal oxygen substitution improved the 6MWD compared to placebo in one clinical trial in PAH patients. Due to the positive results in the treatment of patients with PAH, the initiation of this proof-of-concept study is justified.

DETAILED DESCRIPTION:
Most patients with PAH, except those with congenital heart defects and pulmonary-to-systemic shunts, have minor degrees of hypoxemia at rest and during the night.Current recommendations including the pneumological guidelines for LTOT are based on evidence in patients with chronic obstructive pulmonary disease, as data for patients with PH are lacking: When O2 partial pressure is repeatedly <8 kPa (<60 mmHg, alternatively, 90% of O2 saturation), patients are advised to use O2 to achieve a saturation of >8 kPa. The use of ambulatory O2 can be considered when there is evidence of a symptomatic response or correction of exercise-induced desaturation.

There are only few studies investigating the effect of oxygen supply in pulmonary hypertension, most of which merely investigate acute effects of O2 administration. Short-term oxygen administration has been shown to reduce mean pulmonary arterial pressure, pulmonary vascular resistance and to increase cardiac output in PAH patients. In one study, oxygen supply also reversed the progression of PH in patients with chronic obstructive pulmonary disease (COPD). One recent randomized-controlled trial indicates that O2 given during cardiopulmonary exercise significantly improves maximal work rate and endurance. Furthermore, nocturnal oxygen supply for one week significantly improved 6-minute walking distance in patients with PH, sleep-associated breathing difficulties, exercise performance during the day as well as cardiac repolarisation. Patients with Eisenmenger's syndrome gain little benefit from nocturnal O2 therapy.

Whether these positive effects of O2 supplementation during exercise would translate into long-term improvements of exercise capacity, quality of life, hemodynamics and disease progression is not known to date. Up to now, there are no randomised studies suggesting that long-term O2 therapy is indicated or when it should be initiated.

ELIGIBILITY:
Inclusion Criteria Patients in both groups (n = 20; n=10 each group) with precapillary PH, WHO class I -IV (mPAP ≥ 25 mm Hg, pulmonary arterial occlusion pressure ≤15 mm Hg), who are stable on optimized pharmacological treatment for at least six weeks and who do not suffer from other cardio-pulmonary disease will be recruited if arterial or capillary O2 partial pressure is (<60 mmHg; alternatively, 90% of O2 saturation) at rest and/or during physical activity (O2 partial pressure <60 mmHg pO2 90 % ).

* men and women 18 years of age or older
* patient is diagnosed with Pulmonary Arterial Hypertension (World Health Organization (WHO) Category Group 1 (by the WHO Clinical classification system)), including Idiopathic (IPAH), Heritable PAH (HPAH, Familial PAH), associated PAH (APAH) and CTEPH, with exceptions as noted in exclusion criteria
* patient is willing and able to provide written informed consent
* patient is willing and able to comply with the protocol, including required follow-up visits
* Patients experiencing oxygen desaturations ≤90% (or pO2 below 60 mmHg) at rest and/or oxygen desaturations ≤90% (or pO2 below 60 mmHg) during physical activity
* patient has a stable functional class of PAH with no changes of medication during the last two weeks before inclusion

Exclusion Criteria

* Patient is a female who is pregnant, nursing, or of child bearing potential and is not on a reliable form of birth control
* patient with pulmonary venous hypertension
* significant functional limitation in lung function tests (FEV1 <60%,TLC <60%) and CT morphological signs of pulmonary disease
* significant left heart disease, requiring acute pharmacological or interventional treatment
* unstable conditions requiring pharmacological or other treatment, intensive care or relevant severe concomitant disease
* patient is enrolled, has participated within the last thirty days, or is planning to participate, in a concurrent drug and/or device study during the course of this clinical trial. Co-enrolment in concurrent trials is only allowed with documented pre-approval from the study manager that there is not a concern that co-enrolment could confound the results of this trial.
* patient has been initiated on a new oral or parenteral PAH therapy in the last two weekspatient with a cardiac index (CI) <1.8L/min/m^2
* active smoking Status
* patient with severe resting desaturation (repeatedly SpO2 <80%) or severe exercise-induced desaturation (SpO2 ≤75% for ≥10 minutes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
6-minute Walking distance | Change from baseline to 6 months
  To determine the benefits for PH patients from a long-term oxygen therapy (LTOT) given continuously during ≥16h/day for 12 weeks, measured by improvement of exercise performance assessed by the 6 minute walking distance (6MWD).

SECONDARY OUTCOMES:
Quality of life: physical Summation score; short form health Survey 36 (score from 0-100; higher scores indicating better outcome) | Change from baseline to 6 months
  To investigate effects of oxygen treatment on QoL, physical Summation score measured with SF-36 questionnaire
Quality of life: mental Summation score; short form health Survey 36 (score from 0-100; higher scores indicating better outcome) | Change from baseline to 6 months
  To investigate effects of oxygen treatment on QoL, mental Summation score measured with SF-36 questionnaire
Clinical worsening; frequency and type of clinical worsening events | clinical worsening events from baseline to 6 months
  To assess time to worsening of oxygen saturation and time to clinical worsening
cardiac index in liters per minute per square meter (of body surface area) /(CI) | Change from baseline to 6 months
  Assessment of Cardiac Index during RHC
systolic pulmonary arterial pressure | Change from baseline to 6 months
  Right heart catheterization
mean pulmonary arterial pressure | Change from baseline to 6 months
  Right heart catheterization
pulmonary arterial wedge pressure | Change from baseline to 6 months
  Right heart catheterization
right atrial pressure | Change from baseline to 6 months
  Right heart catheterization
pulmonary vascular resistance (PVR) | Change from baseline to 6 months
  Right heart catheterization
cardiac output and ejection fraction (CO, HZV) | Change from baseline to 6 months
  Right heart catheterization
cardiac index (CI) | Change from baseline to 6 months
  Right heart catheterization
blood gas analysis from pulmonary artery | Change from baseline to 6 months
  central venous saturation
Change in systolic pulmonary arterial pressure | Change from baseline to 6 months
  Echocardiography and Stress Doppler Echocardiography
Echocardiography and Stress Doppler Echocardiography | Change from baseline to 6 months
  right ventricular pump function
Peak oxygen consumption | Change from baseline to 6 months
  Cardiopulmonary exercise testing
Peak oxygen consumption/kg body weight | Change from baseline to 6 months
  Cardiopulmonary exercise testing
oxygen Saturation | Change from baseline to 6 months
  Cardiopulmonary exercise testing
oxygen equivalent | Change from baseline to 6 months
  Cardiopulmonary exercise testing
Cardiopulmonary exercise testing | Change from baseline to 6 months
  carbon dioxide equivalent
Oxygen pulse | Change from baseline to 6 months
  Cardiopulmonary exercise testing
ventilatory threshold | Change from baseline to 6 months
  Cardiopulmonary exercise testing
respiratory reserve | Change from baseline to 6 months
  Cardiopulmonary exercise testing
World Health Organization functional classification | Change from baseline to 6 months
  Functional assessment of pulmonary hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for pulmonary hypertension of the Thoraxclinic at the University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Result] Ulrich S, Hasler ED, Saxer S, Furian M, Muller-Mottet S, Keusch S, Bloch KE. Effect of breathing oxygen-enriched air on exercise performance in patients with precapillary pulmonary hypertension: randomized, sham-controlled cross-over trial. Eur Heart J. 2017 Apr 14;38(15):1159-1168. doi: 10.1093/eurheartj/ehx099. PMID 28329240

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04207593/Prot_SAP_000.pdf